CLINICAL TRIAL: NCT03158545
Title: Efficacy Evaluation of 26 Weeks' Dietary Supplementation With DHA- and EPA-enriched Oils on Cerebral Blood Flow in Healthy Adults
Brief Title: 26 Weeks' Dietary Supplementation With DHA- and EPA-enriched Oils on Cerebral Blood Flow in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Pronova BioPharma (Industry)
Responsible Party: Principal Investigator, Philippa Jackson, Dr., Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 44N4
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Neurovascular Coupling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Olive oil Placebo (Placebo Comparator): 3 x 1 g capsules daily Placebo: olive oil
  Interventions: Dietary Supplement: Olive oil Placebo
- EPA-rich (Active Comparator): 3 x 1 g capsules daily containing EPA-enriched oil
  Interventions: Dietary Supplement: EPA-rich
- DHA-rich (Active Comparator): 3 x 1 g capsules daily containing DHA-enriched oil
  Interventions: Dietary Supplement: DHA-rich

INTERVENTIONS:
Dietary Supplement: Olive oil Placebo — olive oil
  Arms: Olive oil Placebo
Dietary Supplement: EPA-rich — EPA-rich omega-3 oil
  Arms: EPA-rich
Dietary Supplement: DHA-rich — DHA-rich omega-3 oil
  Arms: DHA-rich

SUMMARY:
The purpose of this study is to investigate the effects of EPA- and DHA-enriched omega-3 polyunsaturated fatty acid dietary supplements on cerebral blood flow during a series of cognitive, mathematical subtraction tasks and subjective ratings of task difficulty before and after 26 weeks of supplementation

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 to 49 years inclusive
* Males and females
* Self-report of good health

Exclusion Criteria:

* English is not first language (some of the cognitive tasks have only been validated in native English speakers)
* Habitual consumption of oily fish exceeds one fish meal per week (see Appendix I)
* Habitual consumption of omega-3 dietary supplements in the previous 6 months
* Habitual use of dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total; some supplements that do not impact upon cognitive function e.g. garlic, protein, calcium are allowed. Please check with the research team if you are unsure)
* Are a smoker or consume any nicotine replacement products (e.g. chewing gum, e-cigarettes)
* Food allergies or sensitivities to any of the ingredients contained in the investigational product or any other foodstuff
* Pregnant, trying to get pregnant or breast feeding
* Body Mass Index outside of the range 18-35 kg/m2
* High blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Currently taking blood pressure medication
* Currently taking blood thinning medication (e.g. aspirin, warfarin, heparin)
* Have a respiratory disorder that requires regular medication (Note: participants with asthma who only take their medication occasionally/as required are eligible for this study)
* Have frequent migraines that require medication (more than or equal to 1 per month)
* History or current diagnosis of drug/alcohol abuse
* History of kidney or liver disease, or other severe diseases of the gastrointestinal tract (e.g. iron accumulation, iron utilization disorders, hypercalcaemia, hypercalcaemia), that are likely to interfere with metabolism/absorption/secretion of the product under investigation
* History of neurological or psychiatric illness (excluding depressive illness and anxiety)
* History of head trauma
* Sleep disturbances and/or are taking sleep aid medication
* Blood disorders (e.g. anaemia, haemophilia, thrombocytosis)
* Diagnosis of type I or type II diabetes
* Heart disorder, or vascular illness
* Current diagnosis of depression and/or anxiety
* Over- or under-active thyroid
* Chronic gastrointestinal problems (e.g. Inflammatory Bowel Disease, Irritable Bowel Syndrome, celiac disease)
* Any known active infections
* Diagnosed with syphilis, hepatitis, the Human T - lymphotropic virus or the Human Immunodeficiency Virus
* Current or past breast cancer diagnosis and/or a mastectomy
* Health condition that would prevent fulfilment of the study requirements
* Currently participating in or in the past 4 weeks participated in other clinical or nutrition intervention studies

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow | Participants are assessed pre and post 6 months of supplementation
  Near Infrared Spectroscopy Outcomes for cerebral blood flow measurment

SECONDARY OUTCOMES:
Cognitive Performance | Participants are assessed pre and post 6 months of supplementation
  performance on numerical subtraction tasks
Subjective Task Difficulty | Participants are assessed pre and post 6 months of supplementation
  participants rate how mentally challenging they find the cognitive tasks

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Jackson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patan MJ, Kennedy DO, Husberg C, Hustvedt SO, Calder PC, Khan J, Forster J, Jackson PA. Supplementation with oil rich in eicosapentaenoic acid, but not in docosahexaenoic acid, improves global cognitive function in healthy, young adults: results from randomized controlled trials. Am J Clin Nutr. 2021 Sep 1;114(3):914-924. doi: 10.1093/ajcn/nqab174. PMID 34113957